CLINICAL TRIAL: NCT03568331
Title: A Randomized, Double-Blind, Placebo-Controlled Efficacy Study of The Neurokinin-1 Receptor Antagonist VLY-686 in Patients With Atopic Dermatitis
Brief Title: Evaluating the Effects of Tradipitant vs. Placebo in Atopic Dermatitis (EPIONE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VLY-686-3101; EPIONE (Other: Vanda Pharmaceuticals, Inc.)
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Results first posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-04

CONDITIONS: Atopic Dermatitis
Keywords: Chronic Pruritus; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tradipitant (Experimental)
  Interventions: Drug: Tradipitant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tradipitant — Oral Capsule
  Arms: Tradipitant
Drug: Placebo — Oral Capsule
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to be conducted in the United States in subjects with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-lactating female patients aged 18 - 70 years (inclusive);
* Diagnosed with atopic dermatitis;
* Suffering from chronic pruritus;
* Body Mass Index (BMI) of ≥18 and ≤40 kg/m2

Exclusion Criteria:

* Chronic pruritus due to condition other than atopic dermatitis (AD);
* A positive test for drugs of abuse at the screening or evaluation visits;
* Exposure to any investigational medication in the past 8 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- United States (63):
  - Vanda Investigational Site, Birmingham, Alabama
  - Vanda Investigational Site, Tempe, Arizona
  - Vanda Investigational Site, Encino, California
  - Vanda Investigational Site, Fountain Valley, California
  - Vanda Investigational Site, Fremont, California
  - Vanda Investigational Site, Laguna Hills, California
  - Vanda Investigational Site, Lomita, California
  - Vanda Investigational Site, Long Beach, California
  - Vanda Investigational Site, Los Angeles, California
  - Vanda Investigational Site, San Diego, California
  - Vanda Investigational Site, Santa Monica, California
  - Vanda Investigational Site, Denver, Colorado
  - Vanda Investigational Site, Aventura, Florida
  - Vanda Investigational Site, Clearwater, Florida
  - Vanda Investigational Site, Fort Lauderdale, Florida
  - Vanda Investigational Site, Hialeah, Florida
  - Vanda Investigational Site, Miami, Florida
  - Vanda Investigational Site, Miramar, Florida
  - Vanda Investigational Site, Ormond Beach, Florida
  - Vanda Investigational Site, South Miami, Florida
  - Vanda Investigational Site, Tampa, Florida
  - Vanda Investigational Site, Savannah, Georgia
  - Vanda Investigational Site, Boise, Idaho
  - Vanda Investigational Site, Normal, Illinois
  - Vanda Investigational Site, Skokie, Illinois
  - Vanda Investigational Site, Plainfield, Indiana
  - Vanda Investigational Site, Crowley, Louisiana
  - Vanda Investigational Site, Rockville, Maryland
  - Vanda Investigational Site, Towson, Maryland
  - Vanda Investigational Site, Beverly, Massachusetts
  - Vanda Investigational Site, Brighton, Massachusetts
  - Vanda Investigational Site, Fort Gratiot, Michigan
  - Vanda Investigational Site, Saint Joseph, Missouri
  - Vanda Investigational Site, St Louis, Missouri
  - Vanda Investigational Site, Omaha, Nebraska
  - Vanda Investigational Site, Las Vegas, Nevada
  - Vanda Investigational Site, Berlin, New Jersey
  - Vanda Investigational Site, Verona, New Jersey
  - Vanda Investigational Site, Brooklyn, New York
  - Vanda Investigational Site, New York, New York
  - Vanda Investigational Site, Charlotte, North Carolina
  - Vanda Investigational Site, High Point, North Carolina
  - Vanda Investigational Site, Wilmington, North Carolina
  - Vanda Investigational Site, Cincinnati, Ohio
  - Vanda Investigational Site, Dayton, Ohio
  - Vanda Investigational Site, Oklahoma City, Oklahoma
  - Vanda Investigational Site, Tulsa, Oklahoma
  - Vanda Investigational Site, Philadelphia, Pennsylvania
  - Vanda Investigational Site, Pittsburgh, Pennsylvania
  - Vanda Investigational Site, Johnston, Rhode Island
  - Vanda Investigational Site, North Charleston, South Carolina
  - Vanda Investigational Site, Spartanburg, South Carolina
  - Vanda Investigational Site, Chattanooga, Tennessee
  - Vanda Investigational Site, Nashville, Tennessee
  - Vanda Investigational Site, Dallas, Texas
  - Vanda Investigational Site, Pflugerville, Texas
  - Vanda Investigational Site, San Antonio, Texas
  - Vanda Investigational Site, West Jordan, Utah
  - Vanda Investigational Site, South Burlington, Vermont
  - Vanda Investigational Site, Newport News, Virginia
  - Vanda Investigational Site, Norfolk, Virginia
  - Vanda Investigational Site, Richmond, Virginia
  - Vanda Investigational Site, Spokane, Washington

REFERENCES:
- See also: Study Webpage — https://advandastudy.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tradipitant | Placebo
Started | 188 | 187
Completed | 142 | 144
Not Completed | 46 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tradipitant | Placebo | Total
Number analyzed (Participants) | 188 | 187 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (14.9) | 41.9 (15.1) | 41.8 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 119 | 243
  Male | 64 | 68 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 46 | 88
  Not Hispanic or Latino | 144 | 140 | 284
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 10 | 12 | 22
  Race: Black or African American | 51 | 45 | 96
  Race: Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Race: White | 123 | 123 | 246
  Race: Other | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 188 | 187 | 375
Worst Itch Numeric Rating Scale (NRS) Score [Mean (Standard Deviation); unit: units on a scale] | 8.2 (1.2) | 8.1 (1.3) | 8.2 (1.3)
SCORing Atopic Dermatitis (SCORAD) Index [Mean (Standard Deviation); unit: units on a scale] | 49.56 (14.5) | 50.76 (14.0) | 50.16 (14.3)
Validated Investigator's Global Assessment scale for atopic dermatitis (vIGA-AD) Score [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall due to availability of data.
  Participants
    number analyzed (Participants) | 171 | 170 | 341
    Almost Clear (1) | 2 | 0 | 2
    Mild (2) | 38 | 39 | 77
    Moderate (3) | 113 | 105 | 218
    Severe (4) | 18 | 26 | 44

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Worst Itch in Atopic Dermatitis
Description: Reduction of worst itch in atopic dermatitis as measured by Numerical Rating Scale (NRS). Worst Itch NRS is an assessment tool that is used to report the maximum intensity of participant's itch during a 24-hour recall period. Participants were asked the following question: Please rate the itching severity that describes your worst level of itching in the past 24 hours [0=No Itch, 10=Worst Itch Imaginable].
Time Frame: 8 weeks
Population: All participants randomized (1:1) to placebo or tradipitant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 171 | 170
units on a scale | -3.6 (2.8) | -3.5 (2.75)

2. Secondary Outcome: Improvement of Disease Severity in Atopic Dermatitis
Description: Proportion of participants achieving 50% reduction on the SCORing Atopic Dermatitis (SCORAD) index. SCORAD is an assessment scale used to determine the severity of AD. SCORAD combines the investigator's rating of extent and intensity and the patient reported itch and sleep disturbance. Total score ranges from 0 (absent disease) to 103 (severe disease).
Time Frame: 8 weeks
Population: All participants randomized (1:1) to placebo or tradipitant.
Measure: Count of Participants; unit: Participants
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 171 | 170
Participants | 51 | 54

3. Secondary Outcome: Proportion of Patients With Improvement on Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) of at Least 2-point Reduction
Description: As measured by the validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD). IGA is an assessment scale used to determine severity of AD. It is assessed by the investigator on a 5-point scale (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe) based on erythema, induration/papulation, lichenification, and oozing/crusting.
Time Frame: 8 weeks
Population: All participants randomized (1:1) to placebo or tradipitant.
Measure: Count of Participants; unit: Participants
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 171 | 170
Participants | 37 | 36

4. Post Hoc Outcome: Reduction of Worst Itch in Atopic Dermatitis as Measured by Numerical Rating Scale (NRS), Adjusted for Investigator Global Assessment (IGA)
Description: Worst Itch NRS is an assessment tool that is used to report the maximum intensity of participant's itch during a 24-hour recall period. Participants were asked the following question: Please rate the itching severity that describes your worst level of itching in the past 24 hours [0=No Itch, 10=Worst Itch Imaginable].
Time Frame: 2 weeks
Population: Participants rated 1 or 2 by the IGA, randomized (1:1) to placebo or tradipitant.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 40 | 39
units on a scale | -2.6 [-3.2 to -2.0] | -1.0 [-1.6 to -0.4]

5. Post Hoc Outcome: Reduction in Sleep Disturbances as Measured by SCORing Atopic Dermatitis Index, Adjusted for Investigator Global Assessment
Description: SCORAD is an assessment scale used to determine the severity of AD. SCORAD combines the investigator's rating of extent and intensity and the patient reported itch and sleep disturbance. Total score ranges from 0 (absent disease) to 103 (severe disease).
Time Frame: 2 weeks
Population: Participants rated 1 or 2 by the IGA scale, randomized (1:1) to placebo or tradipitant.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 40 | 39
units on a scale | -2.07 [-2.61 to -1.53] | -0.7 [-1.24 to -0.15]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent up to the final visit (Week 8) regardless of seriousness or relationship to investigational product. Patients with non-serious AEs that are ongoing at the patient's last study visit must be followed until resolution or for 30 days after the patient's last study visit, whichever comes first.
Arm/Group | Tradipitant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/187
Serious Adverse Events (participants affected / at risk) | 2/188 | 1/187
Other Adverse Events (participants affected / at risk) | 23/188 | 11/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tradipitant (N=188) | Placebo (N=187)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tradipitant (N=188) | Placebo (N=187)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 4 (4)
Headache (Nervous system disorders) | 7 (7) | 5 (5)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is restricted from presenting or publishing independently until the expiration of eighteen (18) months from the completion of the Clinical Trial or as otherwise noted in the Investigator's clinical trial agreement.

DOCUMENTS (2):
  • Study Protocol (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT03568331/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT03568331/SAP_001.pdf